CLINICAL TRIAL: NCT02193711
Title: Randomized, Double Blind, Placebo Controlled Trial With Open Label Extension Of Delivra Joint Health Cream In The Treatment Of Pain Caused By Osteoarthritis Of The Knee
Brief Title: Delivra Joint Health Cream In The Treatment Of Pain Caused By Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Delivra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Delivra-001
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Topical Arthritis Cream (Experimental): 1-1.5 ml applied to the skin over the knee in the morning and at bedtime over the entire study period, for a total of 2-3 ml/day.
  Interventions: Other: Topical Arthritis Cream
- Placebo (Placebo Comparator): 1-1.5 ml applied to the skin over the knee in the morning and at bedtime over the entire study period, for a total of 2-3 ml/day.
  Interventions: Other: Topical Arthritis Cream

INTERVENTIONS:
Other: Topical Arthritis Cream
  Other Names: LivRelief Pharmax Rebuild

SUMMARY:
The current clinical trial is designed to test the analgesic and anti-inflammatory efficacy of a topical cream compared to a placebo cream. The study population will be those with mild to moderate osteoarthritis of the knee.

The trial will also provide information about potential side effects and verify the safety of this composition. Blood levels will be done to assess inflammation and to determine whether any systemic absorption has occurred.

Hypothesis/Purpose

* Pain scores after active treatment will be significantly reduced in comparison to placebo.
* There will be an improvement in stiffness and physical function as measured by the WOMAC using the active cream as compared to placebo.
* There will be a decrease in the level of inflammation assessed at baseline, end of week 3 and end of week 6.
* The blood concentration of the active ingredient in the topical cream will not exceed the maximum daily dose that will be consumed by participants.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according to American College of Rheumatology criteria: Knee pain with 3:

  * age >50 years
  * stiffness less than 30 min
  * crepitus,
  * bony tenderness,
  * bony enlargement,
  * no palpable warmth
* Moderate to severe pain, as defined by an average 7-day pain score of greater than 4.0 on an 11-point numerical rating scale for pain intensity (NRS-PI).
* All concurrent medications taken for any reason stable for 14 days
* Ability to follow protocol with reference to cognitive and situational factors (eg. stable housing, ability to attend visits)
* Ability to read and write English
* Willing and able to give informed consent

Exclusion Criteria:

* Currently taking opioids, NSAIDs, warfarin, other anticoagulants, other topical agents for treatment of pain or inflammation
* Allergy to tea tree oil, latex, avocado, soy
* Active conditions such as exzema or psoriasis
* Presence of significant medical disorder that would compromise the participant's safety to take part in the trial (eg. cancer, immunosuppressed)
* Individuals with a history or current disease which may affect the outcome of the trial (ie. Inflammatory, infections joint disease).
* Allergy to plants of the Asteraceae/Compositae/Daisy family.
* Pregnant and breastfeeding women.
* Allergy or other contraindication for acetaminophen use.
* Exercise or transcutaneous electrical nerve stimulation should be excluded prior to and during the trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in mean daily pain diary score from baseline | three weeks
  The primary outcome measure will consist of change in mean daily pain diary score from baseline (average pain score over 7 days pre-treatment) to the final 3 days of the third treatment week. Therefore, the primary analysis is a between group comparison (placebo versus test product) over 3 weeks.

SECONDARY OUTCOMES:
WOMAC | Six weeks
  The Western Ontario and McMaster Universities Arthritis Index is a well validated and widely used measure to assess pain, stiffness and physical function in individuals with OA of the knee or hip. It consists of 24 questions divided into 3 scales (pain, stiffness and physical function). This scale has been found to be sensitive to interventions used for osteoarthritis and is noted by IMMPACT as an example of an appropriate disease specific measure of physical function.
BPI-SF | six weeks
  The BPI pain scale has been widely used and found to provide a reliable and valid measure of pain and pain's interference with physical functioning in seven areas including: general activity, mood, walking ability, work, relations with other people, sleep and enjoyment of life. The instrument consists of a series of 11-point numeric rating scales asking the participant to rate the pain and indicate how much the pain has interfered with seven areas (0 indicating "does not interfere", 10 indicating "completely interferes").
PGIC | six weeks
  The Patient Global Impression of Change Scale (PGIC). This measure is a single-item rating by participants of their improvement with treatment on a 7-point scale that ranges from "very much improved' to "very much worse" with "no-change, as the mid-point.
PGSS | six weeks
  The Patient Global Satisfaction Scale (PGSS) is a 10-point scale with verbal descriptors ranging from "very satisfied" to "not at all satisfied.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CDHA - Pain Management Unit, Halifax, Nova Scotia
  - Canadian College of Naturopathic Medicine, Toronto, Ontario